CLINICAL TRIAL: NCT01826136
Title: Effect of Vibratory Expiratory Pressure on Pulmonary Function After Lung Resection Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YSJeon_Acapella
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Resection Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acapella (Experimental): use of the Acapella device postoperatively
  Interventions: Device: Acapella device
- Control (No Intervention)

INTERVENTIONS:
Device: Acapella device
  Arms: Acapella

SUMMARY:
Postoperative airway clearance and recovery of pulmonary function after lung resection is critical in patients undergoing pulmonary resection surgery. The investigators hypothesized that vibratory positive expiratory pressure using the Acapella device may improve pulmonary function recovery in patients undergoing video-assisted thoracoscopic lung resection surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients between 20 and 65 years old
* undergoing video-assisted thoracoscopic lung resection surgery for suspicious lung cancer
* admission to intensive care unit in extubate state
* with intravenous patient-controlled analgesia

Exclusion Criteria:

* body mass index of less than 15 kg/m2 or more than 30 kg/m2
* history of respiratory tract infection within 3 months
* emergency surgery
* preoperative supplemental oxygen or ventilator care
* preoperative PaO2 of less than 70 mmHg or PaCO2 of more than 50 mmHg
* preoperative FEV1 of less than 30% of predicted value
* unconsciousness or neuromuscular disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
FEV1 on the third postoperative day | 3 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea